CLINICAL TRIAL: NCT06870825
Title: Assessment of Quadriceps Femoris Muscle Function in Patients After Arthroscopic Knee Surgery in Outpatient Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Gintare Repeckaite, assistant teacher, phd student., Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2-BE-2-60/2024
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Meniscus Injury; Meniscus Tear; Arthroscopic Knee Surgeries; ACL Injuries
Keywords: arthroscopic knee surgery; quadriceps femoris atrophy; neuromuscular electrical stimulation; high intensity magnetic field stimulation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-intensity magnetic field muscle stimulation group (Experimental): Group will receive High-intensity magnetic field muscle stimulation group to treat quadriceps muscle atrophy
  Interventions: Device: High-intensity Magnetic Field Muscle Stimulation
- Transcutaneous neuromuscular electrical stimulation group (Active Comparator): Group will receive a Transcutaneous neuromuscular electrical stimulation to treat quadriceps muscle atrophy
  Interventions: Device: Transcutaneous Neuromuscular Electrical Stimulation
- Control group (No Intervention): A Control group, that will receive a standard outpatient rehabilitation plan, without additional quadriceps muscle stimulation methodology.

INTERVENTIONS:
Device: High-intensity Magnetic Field Muscle Stimulation — 1. The procedure is performed for 20 min., 1k/d, 5k/week, a total of 14 times (rehabilitation duration 14 days).
  2. Parameters: applied parameters according to the manufacturer's specified program for muscle stimulation: "muscle strengthening" program
  3. Stimulation site: quadriceps femoris muscle, applied above the motor point approximately 60% of the distance from the upper medial border of the patella to the anterior upper wing of the iliac bone.
  4. device: BLT Super Inductive System
     * Along with muscle stimulation techniques, all subjects will undergo a standardized outpatient rehabilitation plan.
  Arms: High-intensity magnetic field muscle stimulation group
Device: Transcutaneous Neuromuscular Electrical Stimulation — 1. the procedure is performed for 20 min., 1k/d, 5k/week, a total of 14 times (rehab. duration 14 days).
  2. Parameters: applied parameters according to the manufacturer's specified program for muscle stimulation (EMS, P3)
  3. Stimulation site: quadriceps femoris muscle, applied above the motor point.
  4. device: ITO ES-5200
     * Along with muscle stimulation techniques, all subjects will undergo a standardized outpatient rehabilitation plan.
  Arms: Transcutaneous neuromuscular electrical stimulation group

SUMMARY:
The goal of this clinical trial is to learn if a high intensity magnetic field is an effective way to treat quadriceps muscle atrophy after knee arthroscopic surgery in adult patients. The main questions it aims to answer are:

Is high intensity magnetic field muscle stimulation is an effective way to treat quadriceps muscle atrophy Is high intensity magnetic field muscle stimulation is more effective and more tolerable option for quadriceps muscle stimulation than transcutaneous muscle electrical stimulation Researchers will compare high intensity magnetic field muscle stimulation to transcutaneous muscle electrical stimulation and control group, to see if high intensity magnetic field muscle stimulation works to treat quadriceps muscle atrophy.

Participants will:

receive high intensity magnetic field or transcutaneous muscle electrical stimulation 1 time/day for 14 days, Visit the rehabilitation department for testing before/after and 1 month after rehabilitation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of quadriceps muscle stimulation methods: transcutaneous neuromuscular electrostimulation (standard methodology) and high-intensity magnetic field (innovative methodology) stimulation in the rehabilitation of patients after arthroscopic knee surgery, and the impact of the applied methods on the quality of life.

Objectives:

1. To evaluate and check the quadriceps muscle volume, strength, knee joint motion amplitude, pain intensity before and after outpatient rehabilitation and to identify factors that may influence their occurrence.
2. To evaluate and compare the effectiveness of transcutaneous neuromuscular electrical stimulation and high-intensity magnetic field stimulation on changes in quadriceps muscle volume and strength in patients undergoing outpatient rehabilitation after knee joint arthroscopic surgeries.
3. To evaluate the impact of quadriceps muscle size and strength reduction on movement function and quality of life during outpatient rehabilitation, to evaluate changes in condition after outpatient rehabilitation and the previous 1 month, to compare the results obtained.
4. To establish and compare the tolerance of different muscle stimulation methods used and possible adverse reactions after arthroscopic knee joint surgeries.

Subject of the study:

Patients undergoing outpatient rehabilitation, according to the profile of musculoskeletal injuries, 14 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older (working age).
* Arthroscopic knee joint surgery performed
* The dr. orthopedic traumatologist allowed the operated limb to be activated - and rehabilitation to begin
* The period between the operation and the start of rehabilitation is not shorter than 4 weeks and not longer than 2 months.
* Impaired self-service or movement function: Barthel index 80 points or more (according to the order of the Ministry of Health of the Republic of Lithuania) Subjects agreeing to participate in the study

Exclusion Criteria:

* Contraindications to electrostimulation or high-intensity magnetic therapy:

  1. Epilepsy
  2. Implanted electrical devices
  3. Acute rhythm disorders
  4. Oncological diseases (near the stimulation site, active treatment)
  5. Sensory disorders
  6. Skin lesions (near the stimulation site)
  7. Pregnancy.
* Cannot perform the functional tests presented in the study.
* Subjects who cannot be treated with a standardized outpatient rehabilitation plan due to other contraindications (e.g. IC, DVT)
* Subjects who refuse to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Thigh circumference measurement with a centimeter tape (cm) | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  Measuring thigh circumference using a centimeter tape (cm) is a simple yet effective way to track changes in muscle mass, body composition, or to monitor progress. In order to obtain accurate data, the distance between the anterior angle of the iliac wing and the upper edge of the patella is measured with a centimeter tape. Mark the point: ⅓ from the edge of the patella. At the marked point, the thigh circumference is estimated with a centimeter tape, the measurement is repeated 3 times, and the average of the measurements is derived.
Ultrasound assessment of quadriceps muscle cross-sectional area | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  Ultrasound (Mindray DC-80a device) Subject position: During the study, the subject lies on his back, with the knee joints in 15° passive flexion (a cushion is used under the knee joints). During the study, the participants were instructed to relax the thigh muscles. Measurements are performed after the subject has been in a horizontal position for 5 min., to determine the distribution of body fluids [Berg et al., 1993]. Assessment methodology: in order to obtain accurate data, the distance between the greater trochanter of the femur and the upper edge of the patella is measured with a centimeter tape. A point is marked in the distal quarter (75% of the total distance). At the marked point, the ultrasound transducer is placed perpendicular to the longitudinal axis of the thigh on the medial surface, the edge of the quadriceps muscle VM is visualized, and from the starting point, a continuous single image is scanned with the transducer traveling transversely across the thigh along the m
Muscle echogenicity assessed by ultrasound | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  is performed using an ultrasound device (Mindray, DC-80a), in order to obtain accurate data, the distance between the greater trochanter of the femur and the upper edge of the patella is measured with a centimeter tape. A point is marked in the distal quarter (75% of the total distance). At the marked points, the ultrasound transducer is placed perpendicular to the longitudinal axis of the thigh. At the mentioned points, the heads of the quadriceps muscle are visualized, with clear contours, and the image is captured. The image is processed by the ImageJ program, and the visual quantitative scale (VAS echogenicity) is evaluated from 0 to 100.
Muscle strength/power (kg), assessed with a hand-held dynamometer | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  Quadriceps muscle strength will be assessed manually using a manual muscle testing device - Lafayette. Measurements are performed with the subject sitting; the back is supported, the pelvis and knees are bent at an angle of 90°. Then the subjects voluntarily perform 3 consecutive maximal voluntary extensions through the knee joint. (contraction time 3 sec., rest time 7 sec.), the highest value during the assessment was considered the maximal force.
Knee joint pain intensity | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  Pain at rest and during movement will be assessed using the visual analogue scale (VAS)-a line marked with dashes and marked with 11 numbers, from 0 to 10. The subject will be asked to mark a number that indicates the intensity of the pain experienced. Pain is assessed on a scale of 0 to 10, where 0 is no pain, 1, 2, 3 is mild pain, 4, 5, 6 is severe pain, 7, 8, 9 is very severe pain, and 10 is unbearable pain.

SECONDARY OUTCOMES:
Range of motion through the knee joint | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  Active range of motion through the joints is measured with a plastic goniometer (SEAHAN® Grid, 360° per 1° 20 cm) using the neutral zero method. The minimum significant change in range of motion is 5°. The measurements will be repeated three times. After adding all the results obtained during one measurement, the arithmetic mean is calculated.
6-minute walk test | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  The test was used to assess the level of physical fitness. Subjects were asked to walk at their usual maximum pace along a 30-meter long, level, straight hospital corridor without encouragement. The test measured the distance the patient walked in 6 minutes.
Quality of life questionnaire | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  The European Quality of Life and Health Status Questionnaire (EQ-5D-3L) is a standardized quality of life and health status assessment scale developed by the international EuroQoL group. This questionnaire consists of two parts: i. a descriptive part of 5 questions, in which the subject rates his/her health status in 5 dimensions: mobility, self-care, usual activities, pain or discomfort, anxiety or depression, choosing from three options (no problems, some problems or moderate pain, major problems); ii. a visual analogue scale, in which the subject is asked to rate his/her health status on a scale from 0 to 100, where 100 is the highest rating and 0 is the lowest.
Tolerating of interventions | Assessments are performed at the beginning, end, and 1 month after rehabilitation.
  Patients are asked to answer the following questions posed by the researcher:
  1. "Did you experience any discomfort/pain during the procedure?"
  2. "What was the intensity of the discomfort/pain during the stimulation and for the first 2-3 hours after the stimulation" (subjects were asked to rate the pain on the VAS scale)
  3. "Do you have any other comments that are important to you about the discomfort/sensations experienced during the procedure? If so, describe them"

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
For now, we do not have enough human and financial resources to share IPD, but if our circumstances change, we are open to reconsider this decision.